CLINICAL TRIAL: NCT02656134
Title: Small Bowel Endoscopic Evaluation in Familial Adenomatous Polyposis: A Prospective Clinical, Immunopathologic and Molecular Analysis
Brief Title: Small Bowel Endoscopic Evaluation in Familial Adenomatous Polyposis (FAP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Marianny Sulbaran, GI endoscopist, ongoing MSc, PhD, University of Sao Paulo
Other Study IDs: Small bowel profile in FAP
Record Dates: First submitted 2016-01-02; First posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Duodenoscopy; Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Small bowel biopsies and blood samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Duodenoscopy and enteroscopy — All patients will undergo duodenoscopy and classified according to Spigelman. Patients classified as Spigelman III and IV will undergo enteroscopy.
Genetic: Molecular analysis. — DNA analysis
  Other Names: Immunohistochemistry

SUMMARY:
Background and study aim The relative risks of duodenal adenocarcinoma and ampullary carcinoma in Familial Adenomatous Polyposis (FAP) have been estimated 100 to 330 times higher than in general population. However risk factors, including a genotype-phenotype association for duodenal cancer in FAP has not been fully understood. The aim of this study is to determine risk factors associated with the development of advanced duodenal polyposis and ampullary adenomas in colectomized patients with FAP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Familial Adenomatous Polyposis with colectomy, or scheduled for surgery.

Exclusion Criteria:

* Pregnancy, lactation

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Familial Adenomatous Polyposis with colectomy, or scheduled for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Genetic profile in FAP patients | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marianny Sulbaran, MD, Principal Investigator — PhD
Locations (1):
- University of Sao Paulo Medical School, São Paulo, Brazil

REFERENCES:
- [Background] Campos FG, Sulbaran M, Safatle-Ribeiro AV, Martinez CA. Duodenal adenoma surveillance in patients with familial adenomatous polyposis. World J Gastrointest Endosc. 2015 Aug 10;7(10):950-9. doi: 10.4253/wjge.v7.i10.950. PMID 26265988
- [Background] Spigelman AD, Talbot IC, Penna C, Nugent KP, Phillips RK, Costello C, DeCosse JJ. Evidence for adenoma-carcinoma sequence in the duodenum of patients with familial adenomatous polyposis. The Leeds Castle Polyposis Group (Upper Gastrointestinal Committee). J Clin Pathol. 1994 Aug;47(8):709-10. doi: 10.1136/jcp.47.8.709. PMID 7962621
- [Background] Groves CJ, Saunders BP, Spigelman AD, Phillips RK. Duodenal cancer in patients with familial adenomatous polyposis (FAP): results of a 10 year prospective study. Gut. 2002 May;50(5):636-41. doi: 10.1136/gut.50.5.636. PMID 11950808
- [Background] Mathus-Vliegen EM, Boparai KS, Dekker E, van Geloven N. Progression of duodenal adenomatosis in familial adenomatous polyposis: due to ageing of subjects and advances in technology. Fam Cancer. 2011 Sep;10(3):491-9. doi: 10.1007/s10689-011-9433-2. PMID 21416262